CLINICAL TRIAL: NCT00734786
Title: Efficacy and Safety of a Cutaneous Formulation of Gonyautoxin 2/3 (GTX 2/3) for the Treatment of Facial Wrinkles. Study # CLN 08-003.
Brief Title: Efficacy and Safety of a Cutaneous Formulation of Gonyautoxin 2/3 (GTX 2/3) for the Treatment of Facial Wrinkles
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study cancelled.
Sponsor: Phytotox SA (Industry)
Responsible Party: Dra Silvia Pérez Damonte, CLAIM
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CLN 08-003
Record Dates: First submitted 2008-08-07; First posted 2008-08-14 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Facial Wrinkles
Keywords: gonyautoxin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Placebo Comparator): Volunteers will be their own control by randomly receiving the active on one face side and the placebo on the opposite one.
  Interventions: Other: Wrinkle cream application

INTERVENTIONS:
Other: Wrinkle cream application — Single application on the crow's feet wrinkles. Placebo cream will be applied on one side, the active cream on the other side.
  Other Names: No other product will be used.

SUMMARY:
The main objective of the trial is to determine whether the current topical formulation of GTX 2/3 reduces the wrinkling of the skin (crow's feet) after a single application

Other evaluation criteria include: safety assessment and local tolerance, depth of facial wrinkles (video microscopy imaging).

DETAILED DESCRIPTION:
This is a single volunteer group study. Each volunteer will be her own control. A volunteer will receive the active product containing cream on one side of her face and will receive the placebo cream on the other side.

ELIGIBILITY:
Inclusion Criteria:

* Women with no bearing-child potential or with adequate birth control method.
* Volunteers between 30 to 60 years of age.
* Subjects with bilateral crow's feet wrinkles.
* Regular user of cosmetic products, willing and able to comply with the study objectives.
* Signed informed consent.

Exclusion Criteria:

* Any medical condition or any use of a medication that could modify the study results (e.g.: NSAIDs, immunosuppressant drugs, insulin...).
* Any other significant medical condition (e.g.: diabetes mellitus, heart disease, liver disease...).
* Any other condition that in the investigator's opinion could not be appropriate with the participation in this trial.
* Any health condition that could affect the evaluation of study parameters.
* Acute or chronic skin disease.
* History of allergic reaction to cosmetic compounds.
* Pregnancy, planned pregnancy or breast-feeding.
* Allergy to shellfish, fish or sea product (seaweed).
* Known or suspected hypersensitivity to any of the study product compounds.
* Participation in another clinical trial within 30 days previous to enrolment.
* Known or suspected alcohol or drug abuse.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-09 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Depth of facial wrinkles | 24 hours

SECONDARY OUTCOMES:
Local and general tolerance | 1day

CONTACTS AND LOCATIONS:
Overall Officials: Silvia H Pérez-Damonte, PhD, Principal Investigator — CLAIM
Locations (1):
- CLAIM, Buenos Aires, Buenos Aires F.D., Argentina